CLINICAL TRIAL: NCT02005367
Title: Outcome of a Novel Person-Centered Treatment Component for Substance Use Treatment
Brief Title: A Novel Person-Centered Treatment Component for Substance Use Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hampton VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Kathleen Decker, Prinicipal Investigator, Hampton VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-001
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Substance Use Disorders; Depression; Bipolar Disorder; Psychosis; Personality Disorders
Keywords: substance use treatment; person-centered treatment; residential treatment outcomes; dual diagnosis; recovery model; psychosocial treatment
MeSH Terms: conditions — Substance-Related Disorders; Depression; Bipolar Disorder; Psychotic Disorders; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DAP-CP (No Intervention): 512 patients who elected to participate in the Drug Abuse Core Program alone (DAP-CP).
- Natural Recovery-Horticulture (Experimental): Participants in Natural Recovery-Horticulture received a one-hour small group therapy session during the week using one module per week with a staff facilitator and also pursued four hours of their hobby on each weekend day for up to 14 weeks.
  Interventions: Behavioral: Natural Recovery-Horticulture
- Natural Recovery-Art/Music (Experimental): Participants in Natural Recovery-Art/Music received a one-hour small group therapy session during the week using one module per week with a staff facilitator and also pursued four hours of their hobby on each weekend day for up to 14 weeks.
  Interventions: Behavioral: Natural Recovery-Art/Music

INTERVENTIONS:
Behavioral: Natural Recovery-Horticulture — Participants in Natural Recovery-Horticulture received a one-hour small group therapy session during the week using Horticulture modules with a staff facilitator while DAP-CP participants attended a large psychoeducational group at that time.
  Natural Recovery participants also pursued four hours of gardening on each weekend day while DAP-CP attended large-group lectures.
  Arms: Natural Recovery-Horticulture
Behavioral: Natural Recovery-Art/Music — Participants in Natural Recovery-Art/Music received a one-hour small group therapy session during the week using Art/Music modules with a staff facilitator while DAP-CP participants attended a large psychoeducational group at that time. Natural Recovery participants also pursued four hours of art or music on each weekend day while DAP-CP attended large-group lectures.
  Arms: Natural Recovery-Art/Music

SUMMARY:
A person-centered substance use treatment component, the Natural Recovery Program, was developed in a residential substance use treatment setting. The Natural Recovery Program is comprised of small group therapy combined with pursuit of hobbies. The study examined treatment retention, treatment completion and satisfaction of participants of Natural Recovery compared to those who participated in core residential treatment activities alone.

DETAILED DESCRIPTION:
METHODS: Retrospective record review of 643 veterans in an inpatient Mental Health Recovery and Rehabilitation Program was used to determine if participants of Natural Recovery had a different rate of treatment retention and completion than those who participated in the core program alone. Univariate and multivariate analysis was conducted on: participation in the Natural Recovery Program, comorbid psychiatric disorders, legal, medical and psychiatric issues.

PARTICIPANTS: The records of 643 veterans treated in DAP (residential rehabilitation treatment program) at a Veteran's Administration hospital between November, 2009 and March, 2011 were analyzed retrospectively in a quasi-experimental design. The researchers were not blind to participation and participation in the program was an elective component, not randomized. All patients enrolled in DAP were eligible to participate in a novel program called Natural Recovery. Fifteen percent participated in Natural Recovery-Horticulture (n=101), five percent participated in Natural Recovery-Art/Music (n=30) and seventy-nine percent elected to participate in the DAP Core Program only (DAP-CP) (n=512). One percent (n=8) participated in both tracks of Natural Recovery.

PROCEDURE: Participants in Natural Recovery received a one-hour small group therapy session during the week using modules with a staff facilitator while DAP-CP participants attended a large psychoeducational group at that time. Participants in Natural Recovery were given a choice of tracks, either Horticulture or Art/Music based on personal preference. The modules employ analogies between the recovery process and their chosen hobby. Although hobbies were different between the two tracks of Natural Recovery, the fourteen modules covered the same concepts; only the analogy portion of each handout differed.

Natural Recovery participants also pursued four hours of their hobby on each weekend day while DAP-CP participants received large group psychoeducational lectures on weekends during the same amount of time. Thus, total substance use treatment hours between Natural Recovery participants and DAP core program (DAP-CP) participants were equivalent. Additionally, all Natural Recovery-Art/Music, Natural Recovery-Horticulture and DAP-CP participants received one "Leisure Education" lecture.

All participants were free to pursue hobbies during treatment but Natural Recovery participants received materials (access to gardening tools and gardening zones, were provided musical instruments and/or art supplies) to pursue their choice of hobby on the weekend. DAP-CP participants could pursue hobbies during treatment but were not provided musical instruments or art materials, nor did they have access to gardening tools to work in the garden although they could walk in it.

MATERIALS: The modules of Natural Recovery have been previously published and constitute 14 topics, each of which is discussed weekly for 14 weeks [33]. Participants could repeat Natural Recovery modules if their length of stay exceeded 14 weeks. The total number of modules was recorded for each participant.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in the residential substance use treatment program

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Treatment Completion | Up to 150 days
  Treatment completion was defined as regular discharge from the program, which was between 1 and 150 days.

SECONDARY OUTCOMES:
Treatment Retention | up to 150 days
  Treatment retention was defined as the number of days in treatment, from 1-150 days.
Satisfaction with program | up to 150 days
  Satisfaction with either DAP-CP, Natural Recovery-Horticulture or Natural Recovery-Art/Music was measured at the time of discharge on a Likert scale of 1-5 where 5 was highest.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Decker, MD, Principal Investigator — Hampton VAMC
Locations (1):
- Hampton VAMC, Department of Mental Health & Behavioral Sciences, Hampton, Virginia, United States

REFERENCES:
- [Background] Decker, KP: Natural Recovery Program. In Mental Health Residential Rehabilitation Treatment Program (MH RRTP) Promising Practices Compendium: Improving Veterans' Mental Health Care for the 21st Century, Edited by Angela Gerolamo, Jennifer McGovern, Amy Krilla Overcash, Kester St. Kitts, Nikkilyn Morrison, Grace Roemer. Mathematica Policy Research; 2011: p. 24 and p. 184-222.